CLINICAL TRIAL: NCT00048997
Title: A Phase III Comparison Of Prophylactic Cranial Irradiation (PCI) Versus Observation In Patients With Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy in Preventing Central Nervous System (CNS) Metastases in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0214; CDR0000257200; ECOG-RTOG-0214
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic cranial irradiation (PCI) (Experimental): Radiation therapy
  Interventions: Radiation: Radiation therapy
- Observation (Other): Observation
  Interventions: Other: Observation

INTERVENTIONS:
Radiation: Radiation therapy — PCI is given to the whole brain in a dose of 2 Gy per fraction, 5 days per week, for 3 weeks for a total dose of 30 Gy.
  Arms: Prophylactic cranial irradiation (PCI)
Other: Observation
  Arms: Observation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known if giving radiation therapy to the head is effective in preventing CNS metastases in patients who have stage III non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying how well radiation therapy to the head works in preventing CNS metastases in patients who have been previously treated for stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether prophylactic cranial irradiation improves survival after effective locoregional/systemic therapy in patients with stage IIIA or IIIB non-small cell lung cancer.
* Determine the neuropsychologic impact of this therapy in these patients.
* Assess quality of life of patients receiving this therapy.
* Determine the impact of this therapy on the incidence of CNS metastases in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (IIIA vs IIIB), histology (non-squamous cell vs squamous cell), and prior surgery (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo prophylactic cranial irradiation 5 days a week for 3 weeks.
* Arm II: Patients undergo observation.

Patients are followed 3 months during the first year, every 6 months for 2-3 years and then annually thereafter. Quality of life is assessed at baseline and at months 6, 12, 24, 36, and 48.

PROJECTED ACCRUAL: A total of 1,058 patients (529 per treatment arm) will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage IIIA or IIIB non-small cell lung cancer

  * Complete response, partial response, or stable disease after definitive locoregional therapy (with surgery and/or radiation therapy, with or without chemotherapy (chemotherapy alone does not constitute definitive therapy))

    * No more than 16 weeks since prior therapy
* No progressive disease
* No extracranial distant metastatic disease
* No suspicion of CNS metastases by MRI or CT scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other malignancy within the past 3 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic therapy

Chemotherapy

* See Disease Characteristics
* No concurrent anticancer cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior cranial irradiation

Surgery

* See Disease Characteristics

Other

* Recovered from all prior therapies
* No concurrent enrollment on any other phase III study that has progression-free, disease-free, or overall survival as an endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2002-09; Primary Completion 2008-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M. Gore, MD, Study Chair — Medical College of Wisconsin; James A. Bonner, MD, Study Chair — University of Alabama at Birmingham
Locations (14):
- United States (14):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Osborn, Scottsdale, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Resurrection Medical Center, Chicago, Illinois
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - MetroWest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington

REFERENCES:
- [Background] Gondi V, Paulus R, Bruner D, et al.: Prognostic significance of QOL deterioration during early lung cancer survivorship: secondary analysis of RTOG 0212 and 0214. [Abstract] J Clin Oncol 29 (Suppl 15): A-6061, 2011.
- [Result] Gore EM, Bae K, Wong SJ, Sun A, Bonner JA, Schild SE, Gaspar LE, Bogart JA, Werner-Wasik M, Choy H. Phase III comparison of prophylactic cranial irradiation versus observation in patients with locally advanced non-small-cell lung cancer: primary analysis of radiation therapy oncology group study RTOG 0214. J Clin Oncol. 2011 Jan 20;29(3):272-8. doi: 10.1200/JCO.2010.29.1609. Epub 2010 Dec 6. PMID 21135270
- [Result] Sun A, Bae K, Gore EM, Movsas B, Wong SJ, Meyers CA, Bonner JA, Schild SE, Gaspar LE, Bogart JA, Werner-Wasik M, Choy H. Phase III trial of prophylactic cranial irradiation compared with observation in patients with locally advanced non-small-cell lung cancer: neurocognitive and quality-of-life analysis. J Clin Oncol. 2011 Jan 20;29(3):279-86. doi: 10.1200/JCO.2010.29.6053. Epub 2010 Dec 6. PMID 21135267
- [Result] Gore E. RTOG 0214: a phase III comparison of prophylactic cranial irradiation versus observation in patients with locally advanced non-small cell lung cancer. Clin Adv Hematol Oncol. 2005 Aug;3(8):625-6. No abstract available. PMID 16167048
- [Derived] Sun A, Hu C, Wong SJ, Gore E, Videtic G, Dutta S, Suntharalingam M, Chen Y, Gaspar LE, Choy H. Prophylactic Cranial Irradiation vs Observation in Patients With Locally Advanced Non-Small Cell Lung Cancer: A Long-term Update of the NRG Oncology/RTOG 0214 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):847-855. doi: 10.1001/jamaoncol.2018.7220. PMID 30869743

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylactic Cranial Irradiation (PCI): PCI is given to the whole brain in a dose of 2 Gy per fraction, 5 days per week, for 3 weeks for a total dose of 30 Gy.
Period: Overall Study
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Started | 176 | 180
Completed | 163 (Subjects contributing data to the primary analysis are considered to have completed the study.) | 177
Not Completed | 13 | 3
Not completed — Protocol Violation | 7 | 2
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients with consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation | Total
Number analyzed (Participants) | 163 | 177 | 340
Age, Continuous [Median (Full Range); unit: years] | 62 [38 to 81] | 60 [38 to 81] | 61 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 67 | 127
  Male | 103 | 110 | 213

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. This analysis was planned to occur when all patients had been potentially followed for at least 12 months.
Time Frame: From randomization to last follow-up. Analysis occurred after all patients had been on study for at least 12 months. Maximum follow-up at time of analysis was 96 months.
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 163 | 177
months | 28.5 [23.6 to 34.9] | 25.3 [21.0 to 32.2]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; This study was designed to detect a 20% relative improvement in hazard rate: null hypothesis (observation): MST (median survival time) = 23.5 mo.; alternative hypothesis (PCI): MST= 29.4 mo. A one-sided log-rank test at a significance level of 0.025 would have 80% power to detect this difference with a sample size of 1007 patients (527 deaths were required for the final analysis); Test type: Superiority or Other; p = 0.2853, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.84 to 1.38] — Prophylactic cranial irradiation (PCI) is the reference arm for the hazard ratio

2. Secondary Outcome: Percentage of Subjects With Deterioration in the Hopkins Verbal Learning Test - Revised (HVLT-R) Recall Score at One Year
Description: The HVLT-R assesses verbal learning and memory. It incorporates 6 different forms to mitigate practice effects of repeated administrations. Each form includes 12 nouns (targets) with 4 words drawn from 3 semantic categories, which differ across the 6 forms. The recall part of the test involves memorizing a list of 12 targets for 3 consecutive trials for immediate recall. The raw score is derived by summing the number of targets correctly recalled and ranges from 0 to 36 with a higher score indicating better functioning. A patient was classified with deterioration if there was a statistically significant decrease in score from baseline to one year as determined by the method of reliable change index.
Time Frame: Baseline and one year post study entry
Population: All eligible patients with a baseline and 12 month HVLT-R assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 38 | 45
percentage of participants | 26 [13 to 43] | 7 [1 to 18]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; Test type: Superiority; p = 0.01, Z-test, 2-sided; 2-sided significance level = 0.05

3. Secondary Outcome: Percentage of Subjects With Deterioration in the Hopkins Verbal Learning Test - Revised (HVLT-R) Delayed Recall Score at One Year
Description: The HVLT-R assesses verbal learning and memory. It incorporates 6 different forms to mitigate practice effects of repeated administrations. Each form includes 12 nouns (targets) with 4 words drawn from 3 semantic categories, which differ across the 6 forms. The delayed recall part of the test involves memorizing a list of 12 targets and recalling them after a 20-minute delay. The raw score is derived by summing the number of targets correctly recalled and ranges from 0 to 12 with a higher score indicating better functioning. A patient was classified with deterioration if there was a statistically significant decrease in score from baseline to one year as determined by the method of reliable change index.
Time Frame: Baseline and one year post study entry
Population: All eligible patients with a baseline and 12 month HVLT-R assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 31 | 40
percentage of participants | 32 [17 to 51] | 5 [1 to 17]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; Test type: Superiority; p = 0.008, Z-test, 2-sided; Significance level = 0.05

4. Secondary Outcome: Percentage of Subjects With Deterioration in Global Health Status From the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) at One Year
Description: The EORTC QLQ is an integrated system for assessing the health-related quality of life (QOL) of cancer patients participating in international clinical trials. The QLQ Core-30 (QLQ-C30 ) is a 30-item self-report questionnaire that has patients rate the items on a 4-point scale, with 1 "not at all" to 4 "very much" and is composed of both multi-item scales and single-item measures, including 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea and vomiting, pain), a global health status, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). The raw score is calculated as the mean of component items. This score is then standardized such that all of the scales and single-item measures range in score from 0-100. A high score for the global health status represents a high QOL. An increase from baseline to one year by >= 10 points was considered deterioration.
Time Frame: Baseline and one year from randomization
Population: All eligible patients with a baseline and 12 month EORTC QLQ-C30 global health status score
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 37 | 47
percentage of participants | 22 [1 to 38] | 34 [21 to 49]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; Test type: Superiority; p = 0.20, Z-test, 2-sided; Significance level = 0.05

5. Secondary Outcome: Percentage of Subjects With Deterioration in Cognitive Functioning From the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) at One Year
Description: The EORTC QLQ is an integrated system for assessing the health-related quality of life (QOL) of cancer patients participating in international clinical trials. The QLQ Core-30 (QLQ-C30 ) is a 30-item self-report questionnaire that has patients rate the items on a 4-point scale, with 1 "not at all" to 4 "very much" and is composed of both multi-item scales and single-item measures, including 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea and vomiting, pain), a global health status, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). The raw score is calculated as the mean of component items. This score is then standardized such that all of the scales and single-item measures range in score from 0-100. A high score for a functional status represents a high QOL. An increase from baseline to one year by >= 10 points was considered deterioration.
Time Frame: Baseline and one year from randomization
Population: All eligible patients with a baseline and 12 month EORTC QLQ-C30 cognitive functioning score
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 37 | 47
percentage of participants | 41 [25 to 58] | 25 [14 to 40]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; Test type: Superiority; p = 0.14, Z-test, 2-sided; Significance level = 0.05

6. Secondary Outcome: Percentage of Subjects With Deterioration in Fatigue From the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) at One Year
Description: The EORTC QLQ is an integrated system for assessing the health-related quality of life (QOL) of cancer patients participating in international clinical trials. The QLQ Core-30 (QLQ-C30 ) is a 30-item self-report questionnaire that has patients rate the items on a 4-point scale, with 1 "not at all" to 4 "very much" and is composed of both multi-item scales and single-item measures, including 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea and vomiting, pain), a global health status, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). The raw score is calculated as the mean of component items. This score is then standardized such that all of the scales and single-item measures range in score from 0-100. A high score for a symptom scale/item represents a high level of symptomatology/problems. An increase from baseline to one year by >= 10 points was considered deterioration.
Time Frame: Baseline and one year from randomization
Population: All eligible patients with a baseline and 12 month EORTC QLQ-C30 cognitive fatigue score
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 38 | 47
percentage of participants | 34 [20 to 51] | 28 [16 to 43]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; Test type: Superiority; p = 0.52, Z-test, 2-sided; Significance level = 0.05

7. Secondary Outcome: Percentage of Subjects With Deterioration in Future Uncertainty From the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Brain-20 (EORTC QLQ-B20) at One Year
Description: The EORTC QLQ-B20 is a 20-item self-report that assesses 11 symptom scales/items such as future uncertainty, visual disorder, motor dysfunction, and communication deficit. Items are presented as questions on a scale ranging from 1 = "not at all" to 4 = "very much." It is meant for use among brain cancer patients varying in disease stage and treatment modality (i.e. surgery, chemotherapy, radiotherapy, etc.) and should always be complemented by the QLQ-C30. The raw score is calculated as the mean of component items. This score is then standardized such that all of the scales and single-item measures range in score from 0 to 100. A high score for a symptom scale/item represents a high level of symptomatology/problems. An increase from baseline to one year by >= 10 points was considered deterioration.
Time Frame: Baseline and one year from randomization
Population: All eligible patients with a baseline and 12 month EORTC QLQ-B20 future uncertainty score
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 38 | 47
percentage of participants | 16 [6 to 31] | 21 [11 to 36]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; Test type: Superiority; p = 0.51, Z-test, 2-sided; Significance level = 0.05

8. Secondary Outcome: Percentage of Subjects With Deterioration in Communications Deficit From the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Brain-20 (EORTC QLQ-B20) at One Year
Description: as for outcome 7
Time Frame: Baseline and one year from randomization
Population: All eligible patients with a baseline and 12 month EORTC QLQ-B20 communications deficit score
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 38 | 47
percentage of participants | 39 [24 to 57] | 23 [12 to 38]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; Test type: Superiority; p = 0.11, Other [Z-test, 2-sided]; Significance level = 0.05

9. Secondary Outcome: Number of Subjects With Central Nervous System (CNS) Metastases in the First Year
Description: The presence of metastases were determined by computerized tomography (CT) of the brain with and without contrast or by magnetic resonance imaging (MRI) of the brain with and without gadolinium, using the same method that was done prior to study entry.
Time Frame: From randomization to one year (Scans given at 6 and 12 months and additionally at other times within the time frame if clinically indicated.)
Population: Eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Cranial Irradiation (PCI) | Observation
Number analyzed (Participants) | 163 | 177
Participants | 15 | 36
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation (PCI) vs Observation; The development of CNS metastases was assessed using logistic regression modeling comparing presence vs. absence of brain metastases at 1 year; Test type: Superiority; p = 0.005, Regression, Logistic; 2-sided significance level = 0.05; Odds Ratio (OR) = 2.52, 95% CI 2-sided [1.32 to 4.80] — Reference level = PCI arm

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events (AE). Adverse events are compiled for all eligible patients on the prophylactic cranial irradiation arm who received protocol treatment. Adverse events were not collected on the observation arm and therefore that arm is not shown.
Arm/Group | Prophylactic Cranial Irradiation (PCI)
Serious Adverse Events (participants affected / at risk) | 5/163
Other Adverse Events (participants affected / at risk) | 83/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylactic Cranial Irradiation (PCI) (N=163)
Pain-Other (General disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Mood alteration-depression (Psychiatric disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage-Other (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylactic Cranial Irradiation (PCI) (N=163)
Nausea (Gastrointestinal disorders) | 18
Fatigue (lethargy, malaise, asthenia) (General disorders) | 51
Late RT Toxicity: Other: NOS (General disorders) | 27
Late RT Toxicity: Skin: NOS (Injury, poisoning and procedural complications) | 12
Anorexia (Metabolism and nutrition disorders) | 17
Headache (Nervous system disorders) | 14
Late RT Toxicity: Brain: NOS (Nervous system disorders) | 15
Memory loss (Nervous system disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 38

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet accrual goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.